CLINICAL TRIAL: NCT00957710
Title: Slowing Language Decline in Progressive Aphasia Through Language Rehabilitation: Treatment and Neuroimaging Study
Brief Title: Language Treatment for Progressive Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Regina Jokel, clinician scientist, Baycrest
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: REB 09-24
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Primary Progressive Aphasia; Nonfluent Progressive Aphasia; Semantic Dementia
Keywords: progressive aphasia; semantic dementia; neuroimaging; treatment; errorless learning
MeSH Terms: conditions — Aphasia, Primary Progressive; Primary Progressive Nonfluent Aphasia; Frontotemporal Dementia; Aphasia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- langauge therapy (Other): Naming therapy
  Interventions: Behavioral: Errorless learning

INTERVENTIONS:
Behavioral: Errorless learning — Language testing,20 sessions of language therapy, and 2 neuroimaging sessions for participants with progressive aphasia Language testing and 1 imaging session for healthy controls
  Other Names: treatment for anomia

SUMMARY:
Progressive aphasia is characterized by a steady and progressive loss of language skills in the presence of relatively preserved memory, attention, and thinking. The aim of this study is to slow the progression of language decline in progressive aphasia via language therapy. The first goal of this study is to improve naming abilities of individuals with progressive aphasia. This will be accomplished by carrying out an intensive treatment program for anomia. The second goal is to evaluate whether this intense language treatment re-activates affected areas and/or connections within the language network, using functional Magnetic Resonance Imaging (to measure neural activity in specific brain regions) and Diffusion Tensor Imaging tractography (to measure the connectivity between specific brain regions). This is the first study on progressive aphasia addressing both treatment and imaging in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive aphasia
* Native English speaker or fluent in English
* Adequate hearing and vision (not requiring more than +6 diopter correction)
* Willing and able to participate in each phase of the study (including two fMRI sessions)

Exclusion Criteria:

* Contraindications to fMRI (e.g., claustrophobia, pacemaker, ferromagnetic implant)
* Current medical or psychiatric condition affecting cognition (other than progressive aphasia)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of picture naming | 3 months

SECONDARY OUTCOMES:
Changes on neuroimaging | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Regina Jokel, PhD, Principal Investigator — Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Background] Jokel R, Rochon E, Anderson ND. Errorless learning of computer-generated words in a patient with semantic dementia. Neuropsychol Rehabil. 2010 Jan;20(1):16-41. doi: 10.1080/09602010902879859. PMID 19504403
- [Background] Jokel R, Rochon E, Leonard C. Treating anomia in semantic dementia: improvement, maintenance, or both? Neuropsychol Rehabil. 2006 Jun;16(3):241-56. doi: 10.1080/09602010500176757. PMID 16835150
- [Background] Jokel R, Rochon E, Leonard C. Therapy for anomia in semantic dementia. Brain Cogn. 2002 Jul;49(2):241-4. PMID 15259401
- [Background] Jokel R, Cupit J, Rochon E, Leonard C. Relearning lost vocabulary in nonfluent progressive aphasia with Mosstalk Words. Aphasiology 23(2): 175-191, 2009